CLINICAL TRIAL: NCT05895045
Title: Yoga for Treatment of Overactive Bladder in Pediatric Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00112833
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder; Overactive Bladder Syndrome; Overactive Detrusor
Keywords: bladder; overactive; detrusor; pediatric
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The study will start with two treatment arms. Arm 1 will receive standard behavioral modification and possible pharmacologic intervention for six weeks without other intervention. Arm 2 will receive the same therapies in addition to participating in a weekly yoga session for six weeks. At six weeks, arms 1 and 2 we will switch intervention - Arm 1 will then initiate a weekly yoga session for six weeks with emphasis on the pelvic floor relaxation while Arm 2 will continue with standard behavioral / pharmacologic therapy.
  Patients will be divided into two separate yoga groups based on age. The first group will be comprised of 8-12-year-old and the second group will be comprised of 13 - 18-year-old. These will be divided within each treatment arm (i.e Arm 1.1 and 1.2) and the interventions will remain the same.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1.1: 8-12 yoga first (Experimental)
  Interventions: Behavioral: Yoga
- 1.2: 13-18 yoga first (Experimental)
  Interventions: Behavioral: Yoga
- 2.1: 8-12 yoga second (Experimental)
  Interventions: Behavioral: Yoga
- 2.2: 13-18 yoga second (Experimental)
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — Restorative Vinyasa Yoga

SUMMARY:
The goal of this pilot study is to assess the impact of yoga as a treatment modality in pediatric patients age 8-18 diagnosed with idiopathic overactive bladder as measured by validated questionnaires and urinary biomarkers. The main question it aims to answer is: Does yoga help improve overactive bladder symptoms in this patient population? Participants will take part in a weekly yoga session for a total of 6 weeks with validated questionnaires and urinary samples for biomarkers to be completed at the beginning, middle and end of the study. This study will follow a cross-over study design and patients will receive standard of care while not in the active treatment arm.

DETAILED DESCRIPTION:
Detrusor overactivity, otherwise known as overactive bladder (OAB) is the most common disease of voiding dysfunction in children and is characterized by urgency with or without incontinence. Current understanding of OAB suggests that it is a component of central sensitization whereby the central nervous system is in a persistent state of high reactivity. In this state, patients have lower thresholds for pain and for normal physiologic signals such as the sensation of bladder fullness. Yoga has been shown to favor parasympathetic output and appears to be effective in reversing central sensitization for patients with chronic pain. Further, both central sensitization and OAB have been associated with inflammation and so observation of urinary markers of inflammation allow an objective measurement, along with subjective symptom reporting, to measure treatment effects. Children with OAB are likely to become adults with similar urinary complaints and are also more likely to have anxiety, depression and other problems throughout development and maturation. Treatment for OAB in children is comprised of first conservative management with behavioral therapies including biofeedback, subsequent addition of pharmacologic treatment options and finally more invasive therapies including intradetrusor botulinum toxin injections and neuromodulation.

Yoga has been shown to have some positive health benefits in pediatric patients with pulmonary dysfunction, epilepsy, anxiety/depression and even in pediatric oncology patients with regards to quality of life during treatment. Additionally, yoga has been assessed as an adjunctive therapy for the treatment of urinary incontinence and overactive bladder in predominantly adult female populations. That said, to date there have been no studies assessing the impact of yoga on detrusor overactivity in pediatric patient populations (< 19 years old). This is a pilot study in which the investigators hypothesize that yoga will lead to improved quality of life, reduced urinary symptoms and reduced expression of inflammatory urinary biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years of age
* History of non-neurogenic overactive bladder or detrusor overactivity and/or urinary incontinence (ICD 10 codes respectively - N32.81, N39.498)
* Obtained legally effective informed consent and Health Insurance Portability and Accountability Act (HIPPA) authorization from the participant or the participant's parent/legal guardian
* Minor participant is willing and able to provide assent (as applicable)
* Vancouver Dysfunctional Elimination Syndrome[15] score of ≥11 and a positive modified bother score within 30 days of consent

Exclusion Criteria:

* Known or apparent untreated anatomical abnormality of lower urinary tract (i.e. untreated ureterocele)
* Known neurogenic bladder (e.g., spina bifida, history of spinal cord injury, tethered cord)
* Nerve damage that may impact pelvic floor function
* History of chemodenervation of the bladder (e.g., via intravesical instillation or intradetrusor injection of botulinum toxin)
* Active, untreated UTI at the time of enrollment (UTI undergoing active treatment is allowable)
* Current or previous pregnancy at screening or planned pregnancy during the duration of the study, for females of childbearing potential
* Any condition that, in the judgment of the investigator or treating clinician, precludes participation because it could affect participant safety

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in overactive bladder symptoms | 0, 6 and 12 weeks
  Measured via Vancouver symptom score for Dysfunctional Elimination Syndrome with modified bother score (both parts of same survey assessment to be filled out). VDES score ranging from 5-65 with higher number representing worse symptoms; modified bother score ranges from 1-4 with 1= never bothered and 4= always bothered
Change in expression of nerve growth factor | 0, 6 and 12 weeks
  nerve growth factor urinary biomarker via urine specimen collection
Change in expression of interleukin - 1B | 0, 6 and 12 weeks
  Interleukin-1B urinary biomarker via urine specimen collection
Change in expression of tumor necrosis factor-alpha | 0, 6 and 12 weeks
  tumor necrosis factor-alpha urinary biomarker via urine specimen collection

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No